CLINICAL TRIAL: NCT01609582
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate Cardiovascular Outcomes of TAK-875, 50 mg in Addition to Standard of Care in Subjects With Type 2 Diabetes and With Cardiovascular Disease or Multiple Risk Factors for Cardiovascular Events
Brief Title: Study of TAK-875 in Adults With Type 2 Diabetes and Cardiovascular Disease or Risk Factors for Cardiovascular Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to potential concerns about liver safety (See Detailed Description)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-875_306; 2011-001732-37 (EudraCT Number); U1111-1129-7824 (Registry Identifier: WHO); TAK-875_306CTIL (Registry Identifier: Israel MOH); DOH-27-0313-4117 (Registry Identifier: SANCTR); 12/SC/0504 (Registry Identifier: NRES); NMRR-12-433-12087 (Registry Identifier: NMRR (Malaysia)); PHRR130916-000119 (Registry Identifier: PHRR (Philippines)); 1015031332 (Registry Identifier: TCTIN)
Record Dates: First submitted 2012-05-29; First posted 2012-06-01 (Estimated); Results first posted 2015-08-21 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Type 2 Diabetes; Cardiovascular Disease
Keywords: Drug therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — TAK-875

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAK-875 50 mg (Experimental): TAK-875 50 mg tablets, orally, once daily for up to 6 years.
  Interventions: Drug: TAK-875
- Placebo (Placebo Comparator): TAK-875 placebo-matching tablets, orally, once daily for up to 6 years.
  Interventions: Drug: TAK-875 Placebo

INTERVENTIONS:
Drug: TAK-875 — TAK-875 tablets
  Arms: TAK-875 50 mg
Drug: TAK-875 Placebo — TAK-875 placebo-matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate no excess risk of cardiovascular (CV) composite events exists following long term treatment with TAK-875 compared with placebo.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-875. TAK-875 is being tested to treat people who have diabetes. This study will look at the number of cardiovascular events (for example, heart attacks) of people who take TAK-875 in comparison to placebo in addition to standard care.

The study will enroll approximately 5000 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* TAK-875 50 mg.
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient.

All participants will be asked to take one tablet at the same time each day throughout the study. All participants will be asked to record any time they have low blood sugar symptoms in a diary.

This multi-centre trial will be conducted worldwide, in approximately 700 sites. The overall time to participate in this study is 6 years. Participants will make up to approximately 24 visits to the clinic, with telephone visits conducted on an alternate 6 month schedule starting from Month 27.

Due to potential concerns about liver safety, on balance, the benefits of treating patients with fasiglifam (TAK-875) do not outweigh the potential risks.

For this reason, Takeda has decided voluntarily to terminate the development activities for fasiglifam.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the patient is capable of understanding and complying with protocol requirements, including scheduled clinic appointments.
2. The patient or, when applicable, the patient's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has a diagnosis of type 2 diabetes mellitus.
4. Has an glycosylated hemoglobin (HbA1c) level between 7.0% and 10.5%, inclusive, at Screening. HbA1c testing may be repeated once during Screening.
5. Meets at least one (1) of the following three (3) High Risk Categories (a-c ):

   1. A documented history of myocardial infarction (MI) occurring no less than 2 months (60 days) and no greater than 24 months prior to Screening.
   2. Documented symptomatic peripheral arterial disease (PAD) (at least one (1) of the following three (3) criteria must be satisfied): i) Current intermittent claudication together with documented ankle-brachial index ≤0.85. ii) History of previous vascular intervention for intermittent claudication or resting limb ischemia (example: amputation for arterial disease, peripheral bypass, or history of angioplasty/stenting). iii) History of symptomatic carotid artery disease (requiring revascularization with carotid endarterectomy (CEA) or stenting).
   3. Documented cerebrovascular disease (at least one (1) of the following two (2) criteria must be satisfied): i) A history of transient ischemic attack (TIA) confirmed by a neurologist no greater than 24 months prior to screening and clinically and neurologically stable at randomization. ii) A history of ischemic stroke (IS) (with a Modified Rankin Scale Score ≤3 documented prior to Randomization) not less than 2 months (60 days) and no greater than 24 months prior to Screening, and clinically and neurologically stable at Randomization. The Modified Rankin Scale is located in appendix in protocol.

      Or meets at least one (1) of the following five (5) Intermediate Risk Categories (d-h):
   4. Stable angina with coronary disease documented by the presence of inducible ischemia or scar by stress myocardial perfusion imaging (MPI), echocardiogram or magnetic resonance imaging (MRI) in the past 24 months.
   5. Multi vessel coronary disease, based on coronary angiography, with or without angina, documented by >50% diameter stenosis in at least 2 of the 3 major coronary distributions.
   6. A history of percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) at least 2 months prior to Screening.
   7. The subject has diabetic nephropathy plus (2) of the clinical criteria listed below (i. to vi.). Diabetic nephropathy is defined as either urinary albumin excretion ≥ 30 µg/mg creatinine (3.4 mg/mmol creatinine) (based on a random spot collection) or urinary albumin excretion ≥ 30 mg/24h (based on a 24 h or timed collection). Results must be confirmed on at least two specimens collected within 12 months prior to Screening and no more than 6 months apart: i)Duration of diabetes ≥ 10 years on pharmacological treatment documented within medical records. ii) Confirmed systolic blood pressure (SBP) ≥150 mm Hg on 2 separate days during Screening despite treatment with at least 2 anti-hypertensive medications administered at doses considered optimal by local standard of care. iii) Presence of dyslipidemia as defined by any one (1) of the following confirmed at screening: A. Low density lipoprotein (LDL) > 100 mg/dl (2.59 mmol/L) while on statin therapy administered at maximum tolerated dose or optimal dose based on local standard of care for at least 4 weeks prior to screening. B. LDL > 130 mg/dL (3.37 mmol/L) when not on statin therapy. C. High density lipoprotein (HDL) < 40 mg/dL (1.04 mmol/L) in males or < 45 mg/dL (1.17 mmol/L) in females. D. Fasting Triglyceride >200 mg/dL(2.26 mmol/L). iv) Currently smoking >10 cigarettes per day at Screening. v) Male ≥65 years of age or female ≥70 years of age. vi) Highly selective C-reactive protein (hs-CRP) > 2.0 mg/L in the absence of intercurrent infection or acute process.

   h.) The subject meets at least five (5) of the following clinical criteria: i.) Duration of diabetes ≥10 years on pharmacological treatment documented within medical records. ii) Confirmed systolic blood pressure (SBP) ≥150 mm Hg on 2 separate days during Screening despite treatment with at least 2 anti-hypertensive medications administered at doses considered optimal by local standard of care. iii) Presence of dyslipidemia as defined by any one (1) of the following confirmed at screening: A. Low density lipoprotein (LDL) > 100 mg/dl (2.59 mmol/L) while on statin therapy administered at maximum tolerated dose or optimal dose based on local standard of care for at least 4 weeks prior to screening. B. LDL > 130 mg/dL (3.37 mmol/L) when not on statin therapy. C. High density lipoprotein (HDL) < 40 mg/dL (1.04 mmol/L) in males or < 45 mg/dL (1.17 mmol/L) in females. D. Fasting Triglyceride >200 mg/dL(2.26 mmol/L). iv) Currently smoking >10 cigarettes per day at Screening. v) Male ≥65 years of age or female ≥70 years of age. vi) Highly selective C-reactive protein (hs-CRP) > 2.0 mg/L in the absence of intercurrent infection or acute process.
6. Is able and willing to monitor glucose with a home glucose monitor and consistently record his or her own blood glucose concentrations in patient diaries.
7. A female of childbearing potential who is sexually active with a non-sterilized male partner agrees to routinely use adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after the last dose of study drug.
8. Subjects with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤3x upper limit of normal (ULN) and if ALT or AST elevated above ULN, have chronic, well-compensated liver disease documented by usual clinical parameters.

Exclusion Criteria:

1. Has received any investigational medication within 30 days prior to Screening or any investigational antidiabetic medication or excluded medications within 3 months prior to Screening.
2. Has been randomized into a previous TAK-875 study.
3. Is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, biological or legally adopted child, or sibling) or may consent under duress
4. Is diagnosed with type 1 diabetes mellitus or latent autoimmune diabetes in adults.
5. Is hemodynamically unstable, including severe heart failure (New York Heart Association Class IV) at Screening.
6. Is hospitalized at the Screening Visit for the event associated with the CV inclusion criteria. (Patients who have been discharged from an acute hospital to a cardiac rehabilitation center or nursing home at the time of the Screening Visit or Randomization Visit are not excluded).
7. Has ALT and/or AST levels >3.0x ULN at Screening.
8. Has a total bilirubin level >ULN at Screening. Exception: if a patient has documented Gilbert's Syndrome, the patient will be allowed with an elevated bilirubin level per the investigator's discretion.
9. Has an glomerular filtration rate (estimated) (eGFR) ≤ 15 mL/min/1.73m2 based on Modification of Diet in Renal Disease (MDRD) calculation at Screening and is currently on dialysis or expected to start dialysis within the next 6 months.
10. Has uncontrolled thyroid disease, as determined by the investigator and/or clinical investigation.
11. Has a known history of infection with human immunodeficiency virus (HIV).
12. Has a known active infection with Hepatitis B virus (HBV), or Hepatitis C virus (HCV) requiring antiviral treatment.
13. Has a history of drug abuse (defined as illicit drug use) or a history of alcohol abuse within 2 years prior to Screening.
14. Has any major illness or condition that, in the investigator's opinion, prohibits the patient from participating in the study or meeting the planned visit schedule.
15. Has a history of hypersensitivity, allergies, or has had an anaphylactic reaction(s) to TAK-875.
16. If female, is pregnant (confirmed by laboratory testing, ie, serum or urine human chorionic gonadotropin (hCG), in females of childbearing potential) or lactating or intending to become pregnant before, during, or within 30 days after participating in this study; or intending to donate ova during such time period.
17. Is unable to understand verbal or written English or any other language for which a certified translation of the approved informed consent is available.
18. Has a history of cancer that has been in remission for <5 years prior to Screening. A history of basal cell carcinoma or Stage 1 squamous cell carcinoma of the skin is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3207 (Actual)
Dates: Start 2012-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Medical Director Clinical Science, Study Director — Takeda
Locations (584):
- United States (218):
  - Birmingham, Alabama
  - Dothan, Alabama
  - Mobile, Alabama
  - Muscle Shoals, Alabama
  - Pell City, Alabama
  - Goodyear, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - El Cajon, California
  - Fresno, California
  - Fullerton, California
  - La Mesa, California
  - Laguna Hills, California
  - Los Angeles, California
  - Mission Hills, California
  - National City, California
  - Newport Beach, California
  - Orange, California
  - Paramount, California
  - Pismo Beach, California
  - Redondo Beach, California
  - San Diego, California
  - San Francisco, California
  - San Franciso, California
  - Stockton, California
  - Thousand Oaks, California
  - Torrance, California
  - Valley Village, California
  - Westlake Village, California
  - Denver, Colorado
  - Lakewood, Colorado
  - Bridgeport, Connecticut
  - Danbury, Connecticut
  - Seaford, Delaware
  - Washington D.C., District of Columbia
  - Boynton Beach, Florida
  - Brandon, Florida
  - Chipley, Florida
  - Clearwater, Florida
  - Cocoa, Florida
  - Coral Gables, Florida
  - Coral Springs, Florida
  - Crystal River, Florida
  - Delray Beach, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Inverness, Florida
  - Jacksonville, Florida
  - Jacksonville Beach, Florida
  - Melbourne, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - Ocala, Florida
  - Oviedo, Florida
  - Pembroke Pines, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Trinity, Florida
  - Vero Bearch, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Calhoun, Georgia
  - Conyers, Georgia
  - Cumming, Georgia
  - Norcross, Georgia
  - Roswell, Georgia
  - Suwanee, Georgia
  - Woodstock, Georgia
  - Chicago, Illinois
  - LaGrange, Illinois
  - Springfield, Illinois
  - Anderson, Indiana
  - Avon, Indiana
  - Elkhart, Indiana
  - Greenfield, Indiana
  - Indianapolis, Indiana
  - Muncie, Indiana
  - Ames, Iowa
  - Council Bluffs, Iowa
  - Waterloo, Iowa
  - Augusta, Kansas
  - Hutchinson, Kansas
  - Newton, Kansas
  - Topeka, Kansas
  - Wichita, Kansas
  - Elizabethtown, Kentucky
  - Marrero, Louisiana
  - Monroe, Louisiana
  - Natchitoches, Louisiana
  - New Orleans, Louisiana
  - Sherveport, Louisiana
  - Portland, Maine
  - Annapolis, Maryland
  - Balitmore, Maryland
  - Baltimore, Maryland
  - Fall River, Massachusetts
  - Hyannis, Massachusetts
  - Natick, Massachusetts
  - Springfield, Massachusetts
  - Bay City, Michigan
  - Cadillac, Michigan
  - Flint, Michigan
  - Kalamazoo, Michigan
  - Mount Clemens, Michigan
  - Novi, Michigan
  - Pontiac, Michigan
  - Saginaw, Michigan
  - Troy, Michigan
  - Baxter, Minnesota
  - Saint Cloud, Minnesota
  - Saint Paul, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Nashua, New Hampshire
  - Bridgewater, New Jersey
  - Elizabeth, New Jersey
  - Haddon Heights, New Jersey
  - Linden, New Jersey
  - Mine Hill, New Jersey
  - Somerset, New Jersey
  - South Plainfield, New Jersey
  - Toms Rivers, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Buffalo, New York
  - Mineola, New York
  - New York, New York
  - Saratoga Springs, New York
  - Smithtown, New York
  - Syracuse, New York
  - Burlington, North Carolina
  - Calabash, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Lenoir, North Carolina
  - Mooresville, North Carolina
  - Morganton, North Carolina
  - Raleigh, North Carolina
  - Rocky Mount, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Fairview Park, Ohio
  - Gallipolis, Ohio
  - Kettering, Ohio
  - Marion, Ohio
  - Middleburg Heights, Ohio
  - Perrysburg, Ohio
  - Springfield, Ohio
  - Toledo, Ohio
  - Willoughby Hills, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Chambersburg, Pennsylvania
  - Hanleysville, Pennsylvania
  - Harleysville, Pennsylvania
  - Levittown, Pennsylvania
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Philadelphi, Pennsylvania
  - Scotland, Pennsylvania
  - Uniontown, Pennsylvania
  - East Providence, Rhode Island
  - Pawtucket, Rhode Island
  - Columbia, South Carolina
  - Greer, South Carolina
  - Laurens, South Carolina
  - Simpsonville, South Carolina
  - Bristol, Tennessee
  - Crossville, Tennessee
  - Jackson, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Oak Ridge, Tennessee
  - Tullahoma, Tennessee
  - Austin, Texas
  - Carrollton, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Irving, Texas
  - Katy, Texas
  - Midland, Texas
  - Odessa, Texas
  - Pearland, Texas
  - San Antonio, Texas
  - Spring, Texas
  - Tomball, Texas
  - Victoria, Texas
  - Bountiful, Utah
  - Layton, Utah
  - Salt Lake City, Utah
  - Alexandria, Virginia
  - Danville, Virginia
  - Falls Church, Virginia
  - Hampton, Virginia
  - Manassas, Virginia
  - Wenatchee, Washington
  - Huntington, West Virginia
  - Lewisburg, West Virginia
  - La Crosse, Wisconsin
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
  - Wauwatosa, Wisconsin
- Argentina (27):
  - Bahía Blanca, Buenos Aires
  - Haedo, Buenos Aires
  - La Plata, Buenos Aires
  - Loma Hermosa, Buenos Aires
  - Mar del Plata, Buenos Aires
  - Quilmes, Buenos Aires
  - San Nicolás de los Arroyos, Buenos Aires
  - Zárate, Buenos Aires
  - Trelew, Chubut Province
  - Buenos Aires, Ciudad Autonoma Buenos Aires
  - Ciudad Autonoma Buenos Aires, Ciudad Autonoma Buenos Aires
  - Corrientes, Corrientes Province
  - Córdoba, Córdoba Province
  - Villa Cabrera, Córdoba Province
  - Villa María, Córdoba Province
  - San Salvador de Jujuy, Jujy
  - Godoy Cruz, Mendoza Province
  - Mendoza, Mendoza Province
  - Cipolletti, Río Negro Province
  - Salta, Salta Province
  - Rosario, Santa Fe Province
  - Santa Fe, Santa Fe Province
  - Venado Tuerto, Santa Fe Province
  - Santiago del Estero, Santiago del Estero Province
  - San Miguel de Tucumán, Tucumán Province
  - Córdoba
  - Rosario
- Australia (21):
  - Bruce, Australian Capital Territory
  - Canberra, Australian Capital Territory
  - Garran, Australian Capital Territory
  - Westmead, New South Wales
  - Wollongong, New South Wales
  - Brisbane, Queensland
  - Meadowbrook, Queensland
  - Milton, Queensland
  - Townsville, Queensland
  - Woolloongabba, Queensland
  - Adelaide, South Australia
  - Daw Park, South Australia
  - Elizabeth Vale, South Australia
  - Clayton, Victoria
  - Fitzroy, Victoria
  - Geelong, Victoria
  - Melbourne, Victoria
  - Sale, Victoria
  - Joondalup, Western Australia
  - Bruce
  - Garran
- Brazil (14):
  - Fortaleza, Ceará
  - Brasília, Federal District
  - Goiânia, Goiás
  - Campina Grande do Sul, Paraná
  - Curitiba, Paraná
  - Belém, Pará
  - Recife, Pernambuco
  - Canoas, Rio Grande do Sul
  - Caxias do Sul, Rio Grande do Sul
  - Passo Fundo, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Santa Maria, Rio Grande do Sul
  - Marília, São Paulo
  - São Paulo, São Paulo
- Bulgaria (9):
  - Blagoevgrad
  - Byala
  - Kazanlak
  - Pazardzhik
  - Plovdiv
  - Sevlievo
  - Sofia
  - Stara Zagora
  - Varna
- Canada (21):
  - Calgary, Alberta
  - Spruce Grove, Alberta
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Brampton, Ontario
  - Etobicoke, Ontario
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - Markham, Ontario
  - Oakville, Ontario
  - Ottawa, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Gatineau, Quebec
  - Laval, Quebec
  - Longueuil, Quebec
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Saint-Jérôme, Quebec
  - Saint-Laurent, Quebec
- Croatia (12):
  - Čakovec
  - Karlovac
  - Koprivnica
  - Krapinske Toplice
  - Osijek
  - Rijeka
  - Sisak
  - Slavonski Brod
  - Split
  - Virovitica
  - Zadar
  - Zagreb
- Czechia (15):
  - Choceň
  - České Budějovice
  - Jindřichův Hradec
  - Kroměříž
  - Mariánské Lázně
  - Moravský Krumlov
  - Olomouc
  - Ostrava
  - Ostrava - Moravska Ostrava
  - Ostrava - Vitkovice
  - Prague
  - Praha 4 - Krc
  - Slaný
  - Trutnov
  - Ústí nad Labem
- Estonia (3):
  - Paide
  - Tallinn
  - Tartu
- France (7):
  - Corbeil Essonne, Essonne
  - Corbeil-Essonnes, Essonne
  - Pessac, Gironde
  - Nanterre, Hauts de Seine
  - Nantes, Loire Atlantique
  - Paris, Paris
  - Pierre-Bénite, Rhone
- Germany (14):
  - Friedrichstal, Baden-Wurttemberg
  - Falkensee, Brandenburg
  - Hamburg, Hamburg
  - Kelkheim, Hesse
  - Cologne, North Rhine-Westphalia
  - Dortmund, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Goch, North Rhine-Westphalia
  - Kamp-Lintfort, North Rhine-Westphalia
  - Bad Kreuznach, Rhineland-Palatinate
  - Dippoldiswalde, Saxony
  - Dresden, Saxony
  - Hohenmölsen, Saxony-Anhalt
  - Berlin, State of Berlin
- Hong Kong (2):
  - Hong Kong
  - New Territories
- Hungary (20):
  - Baja
  - Balatonfüred
  - Budaörs
  - Budapest
  - Debrecen
  - Eger
  - Gödöllő
  - Gyula
  - Kecskemét
  - Kistelek
  - Komárom
  - Makó
  - Pécs
  - Szeged
  - Szekszárd
  - Szikszó
  - Szombathely
  - Úrhida
  - Veszprém
  - Zalaegerszeg
- Israel (13):
  - Ashkelon
  - Beer Yaakov
  - Beersheba
  - Giv‘atayim
  - Hadera
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Raanana
  - Safed
  - Tel Aviv
- Italy (5):
  - Florence, Firenze
  - Milan, Milano
  - San Donato Milanese, Milano
  - Sesto San Giovanni, Milano
  - Pavia, Pavia
- Latvia (7):
  - Daugavpils
  - Jelgava
  - Limbaži
  - Ogre
  - Riga
  - Talsi
  - Valmiera
- Lithuania (3):
  - Alytus
  - Kaunas
  - Klaipėda
- Malaysia (15):
  - Johor Bahru, Johor
  - Alor Star, Kedah
  - Kelantan, Kelantan
  - Kota Bharu, Kelantan
  - Kuala Lumpur, Kuala Lumpur
  - Lembah Pantai, Kuala Lumpur
  - Malacca, Melaka
  - Ipoh, Perak
  - Taiping, Perak
  - Taiping, Perak, Perak
  - Kuala Selangor, Selangor
  - Petaling Jaya, Selangor
  - Terengganu, Terengganu
  - Kuala Selangor
  - Terengganu
- Mexico (22):
  - Aguascalientes, Aguascalientes
  - Tijuana, Baja California Norte
  - Chihuahua City, Chihuahua
  - Torreón, Coahuila
  - Durango, Durango
  - Acapulco de Juárez, Guerrero
  - Pachuca, Hidalgo
  - Guadalajara, Jalisco
  - Zapopan, Jalisco
  - Cuauhtémoc, Mexico City
  - Mexico City, Mexico City
  - Morelia, Michoacán
  - Cuernavaca, Morelos
  - Monterrey, Nuevo Le=n
  - Monterrey, Nuevo León
  - San Luis Potosí City, San Luis Potos
  - Culiacán, Sinaloa
  - Cuautitlán Izcalli, State of Mexico
  - Metepec, State of Mexico
  - Tamaulipas, Tamaulipas
  - Xalapa, Veracruz
  - Mérida, Yucatán
- New Zealand (6):
  - Auckland
  - Christchurch
  - Dunedin
  - Palmerston North
  - Tauranga
  - Wellington
- Peru (7):
  - Callao
  - Cusco
  - Huacho
  - Ica
  - La Libertad
  - Lima
  - Piura
- Philippines (9):
  - Baguio City
  - Cebu City
  - Dasmariñas City, Cavite
  - Davao City
  - Iloilo City
  - Marikina City
  - Quezon City
  - Tarlac City
  - Taytay
- Poland (17):
  - Bialystok
  - Gdansk
  - Gliwice
  - Grodzisk Mazowiecki
  - Kamieniec Ząbkowicki
  - Lodz
  - Lublin
  - Oświęcim
  - Parczew
  - Poznan
  - Puławy
  - Radom
  - Ruda Śląska
  - Rzeszów
  - Warsaw
  - Wroclaw
  - Łęczyca
- Romania (10):
  - Bacau
  - Baia Mare
  - Brasov
  - Bucharest
  - Galati
  - Iași
  - Oradea
  - Ploieşti
  - Târgu Mureş
  - Timișoara
- Russia (11):
  - Arkhangelsk
  - Barnaul
  - Kazan'
  - Kemerovo
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Pushkin
  - Saint Petersburg
  - Saratov
  - Yaroslavl
- Slovakia (13):
  - Bratislava
  - Komárno
  - Košice
  - Levice
  - Lučenec
  - Martin
  - Nitra
  - Nové Mesto nad Váhom
  - Prešov
  - Svidník
  - Šahy
  - Trenčín
  - Žilina
- South Africa (11):
  - Port Elizabeth, Eastern Cape
  - Bloemfontein, Free State
  - Johannesburg, Gauteng
  - Kempton Park, Gauteng
  - Krugersdorp, Gauteng
  - Lenasia, Gauteng
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Cape Town, Western Cape
  - Stellenbosch, Western Cape
  - Worcester, Western Cape
- South Korea (7):
  - Wŏnju, Gangwon-do
  - Seongnam-si, Gyeonggi-do
  - Yangsan, Gyeongsangnam-do
  - Jeonju, Jeollabuk-do
  - Busan
  - Gyeonggi-do
  - Seoul
- Taiwan (6):
  - Douliu
  - Kaohsiung City
  - New Taipei City
  - Taichung
  - Tainan
  - Taipei
- Thailand (10):
  - Bangkoknoi, Bangkok
  - Dusit, Bangkok
  - Patumwan, Bangkok
  - Rachathevi, Bangkok
  - Rajtevi, Bangkok
  - Ratchathewi, Bangkok
  - Muang, Changwat Chiang Rai
  - Muang, Changwat Khon Kaen
  - Muang, Changwat Nakhon Ratchasima
  - Muang, Chiang Mai
- Ukraine (12):
  - Donetsk
  - Kharkiv
  - Kyiv
  - Luhansk
  - Mykolayiv
  - Odesa
  - Poltava
  - Simferopol
  - Ternopil
  - Vinnycia
  - Vinnytsia
  - Zaporizhzhia
- United Kingdom (17):
  - Cardiff, Cardiff
  - Truro, Cornwall
  - Exeter, Devon
  - Plymouth, Devon
  - Torquay, Devon
  - Hull, East Riding of Yorkshire
  - Bexhill-on-Sea, East Sussex
  - Portsmouth, Hampshire
  - Watford, Hertfordshire
  - Gillingham, Kent
  - Thornton-Cleveleys, Lancashire
  - Leicester, Leicestershire
  - Liverpool, Merseyside
  - Harrow, Middlesex
  - Northwood, Middlesex
  - Stoke-on-Trent, Staffordshire
  - Swansea, West Glamorgan

REFERENCES:
- [Derived] Shavadia JS, Sharma A, Gu X, Neaton J, DeLeve L, Holmes D, Home P, Eckel RH, Watkins PB, Granger CB. Determination of fasiglifam-induced liver toxicity: Insights from the data monitoring committee of the fasiglifam clinical trials program. Clin Trials. 2019 Jun;16(3):253-262. doi: 10.1177/1740774519836766. Epub 2019 Mar 18. PMID 30880443
- [Derived] Menon V, Lincoff AM, Nicholls SJ, Jasper S, Wolski K, McGuire DK, Mehta CR, Rosenstock J, Lopez C, Marcinak J, Cao C, Nissen SE; GRAND 306 Investigators. Fasiglifam-Induced Liver Injury in Patients With Type 2 Diabetes: Results of a Randomized Controlled Cardiovascular Outcomes Safety Trial. Diabetes Care. 2018 Dec;41(12):2603-2609. doi: 10.2337/dc18-0755. PMID 30459247

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 469 investigative sites in 31 countries; 192 sites in North America, 175 in the Europe, Middle East, and Africa (EMEA) region (including Russia, Ukraine, Israel, and South Africa), 65 in the Asia Pacific region, and 37 in Latin/South America from 01 June 2012 to 05 May 2014.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus (T2DM) and clinically-evident cardiovascular (CV) disease or multiple risk factors for CV events who were inadequately controlled while receiving the standard of care were enrolled in 1 of 2 treatment groups: placebo; fasiglifam 50 milligram (mg).
Groups:
- Placebo: Fasiglifam placebo-matching tablet, orally, once daily for up to 588 days.
- Fasiglifam 50 mg: Fasiglifam 50 mg, tablet, orally, once daily for up to 582 days.
Period: Overall Study
Arm/Group | Placebo | Fasiglifam 50 mg
Started | 1603 | 1604
Treated | 1603 | 1601
Completed | 0 | 0
Not Completed | 1603 | 1604
Not completed — Adverse Event | 20 | 18
Not completed — Lost to Follow-up | 10 | 10
Not completed — Withdrawal by Subject | 21 | 15
Not completed — Study Terminated by Sponsor | 1543 | 1548
Not completed — Other | 9 | 10
Not completed — Randomized, but not treated | 0 | 3

BASELINE CHARACTERISTICS:
Population: The randomized set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fasiglifam 50 mg | Total
Number analyzed (Participants) | 1603 | 1604 | 3207
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (9.03) | 63.4 (9.20) | 63.7 (9.12)
Age, Customized [Number; unit: participants]
  Less than (<) 65 years | 794 | 851 | 1645
  Greater than or equal to (>=) 65 years | 809 | 753 | 1562
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 543 | 563 | 1106
  Male | 1060 | 1041 | 2101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 150 | 119 | 269
  Not Hispanic or Latino | 446 | 477 | 923
  Unknown or Not Reported | 1007 | 1008 | 2015
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 47 | 41 | 88
  Asian | 199 | 205 | 404
  Native Hawaiian or Other Pacific Islander | 6 | 7 | 13
  Black or African American | 79 | 95 | 174
  White | 1265 | 1246 | 2511
  Multiracial/More than 1 race | 7 | 10 | 17
Height [Mean (Standard Deviation); unit: centimeter (cm)] — For this outcome measure, number of participants evaluable were 1598 and 1597 for each arm, respectively.
  centimeter (cm) | 168.1 (9.84) | 167.6 (10.54) | 167.8 (10.20)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 91.14 (19.832) | 91.40 (21.319) | 91.27 (20.586)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — For this outcome measure, number of participants evaluable were 1598 and 1597 for each arm, respectively.
  kilogram per square meter (kg/m^2) | 32.14 (6.107) | 32.45 (7.497) | 32.30 (6.838)
Glycosylated Hemoglobin (HbA1c) Category [Number; unit: participants]
  <8.5 percent (%) | 988 | 936 | 1924
  >=8.5% | 615 | 668 | 1283
Smoking Classification [Number; unit: participants]
  Never smoked | 667 | 668 | 1335
  Current smoker | 330 | 328 | 658
  Ex-smoker | 606 | 608 | 1214
Duration of Diabetes [Mean (Standard Deviation); unit: years] — For this outcome measure, number of participants evaluable were 1602 and 1602 for each arm, respectively.
  years | 13.583 (8.409) | 13.333 (8.321) | 13.458 (8.365)
Region of Enrollment [Number; unit: participants]
  Argentina | 121 | 121 | 242
  Australia | 34 | 35 | 69
  Bulgaria | 21 | 22 | 43
  Canada | 104 | 107 | 211
  Croatia | 16 | 17 | 33
  Czech Republic | 56 | 56 | 112
  Estonia | 13 | 11 | 24
  France | 3 | 4 | 7
  Germany | 30 | 30 | 60
  Hong Kong | 29 | 29 | 58
  Hungary | 74 | 72 | 146
  Israel | 25 | 26 | 51
  Italy | 3 | 3 | 6
  Korea, Republic of | 29 | 27 | 56
  Latvia | 11 | 11 | 22
  Lithuania | 15 | 15 | 30
  Malaysia | 30 | 31 | 61
  Mexico | 26 | 26 | 52
  New Zealand | 20 | 20 | 40
  Peru | 18 | 17 | 35
  Philippines | 25 | 24 | 49
  Poland | 118 | 118 | 236
  Romania | 5 | 4 | 9
  Russian Federation | 25 | 23 | 48
  Slovakia | 31 | 31 | 62
  South Africa | 10 | 10 | 20
  Taiwan, Province of China | 31 | 31 | 62
  Thailand | 29 | 32 | 61
  Ukraine | 76 | 76 | 152
  United Kingdom | 16 | 16 | 32
  United States | 559 | 559 | 1118

OUTCOME MEASURES:

1. Primary Outcome: Time to First Occurrence of Any Component of Primary Major Adverse Cardiovascular Event (MACE) Composite
Description: The time from randomization to the first occurrences of any event in the primary MACE composite was evaluated using Kaplan-Meier analysis. The primary MACE composite comprised cardiovascular (CV) death, nonfatal myocardial infarction (MI), nonfatal stroke, and hospitalization for unstable angina (with or without revascularization).
Time Frame: Baseline up to end of study (up to Day 588)
Population: Full Analysis Set (FAS) included all randomized participants who had baseline and at least 1 post-baseline assessment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Fasiglifam 50 mg
Number analyzed (Participants) | 1603 | 1604
days | NA [NA to NA] — Median time and corresponding 95% confidence interval could not be reached since very low number of participants (<50%) had event related to any component of primary MACE composite. | NA [NA to NA] — Median time and corresponding 95% confidence interval could not be reached since very low number of participants (<50%) had event related to any component of primary MACE composite.

2. Secondary Outcome: Time to First Occurrence of Any Component of Secondary Major Adverse Cardiovascular Event (MACE) Composite
Description: The time from randomization to the first occurrences of any event in the secondary MACE composite was evaluated using Kaplan-Meier analysis. The secondary MACE composite comprised CV death, nonfatal MI, and nonfatal stroke.
Time Frame: Baseline up to end of study (up to Day 588)
Population: Full Analysis Set (FAS) included all randomized participants who had baseline and at least 1 post-baseline assessment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Fasiglifam 50 mg
Number analyzed (Participants) | 1603 | 1604
days | NA [NA to NA] — Median time and corresponding 95% confidence interval could not be reached since very low number of participants (<50%) had event related to any component of secondary MACE composite. | NA [NA to NA] — Median time and corresponding 95% confidence interval could not be reached since very low number of participants (<50%) had event related to any component of secondary MACE composite.

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 30 days after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Fasiglifam 50 mg
Serious Adverse Events (participants affected / at risk) | 197/1603 | 201/1601
Other Adverse Events (participants affected / at risk) | 427/1603 | 415/1601
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1603) | Fasiglifam 50 mg (N=1601)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Atrioventricular block first degree (Cardiac disorders) | 3 | 3
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 7 | 6
Coronary artery occlusion (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 7 | 12
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 9 | 12
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 4
Cardiogenic shock (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 7 | 9
Angina unstable (Cardiac disorders) | 5 | 7
Myocardial infarction (Cardiac disorders) | 5 | 4
Acute coronary syndrome (Cardiac disorders) | 3 | 3
Myocardial ischaemia (Cardiac disorders) | 4 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 3
Right ventricular failure (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 4
Cardio-respiratory arrest (Cardiac disorders) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2
Pituitary haemorrhage (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 2
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 3
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Pancreatic calcification (Gastrointestinal disorders) | 1 | 0
Medical device pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Device malfunction (General disorders) | 0 | 2
Local swelling (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Chest pain (General disorders) | 6 | 8
Non-cardiac chest pain (General disorders) | 3 | 4
Chest discomfort (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 3
Cholelithiasis (Hepatobiliary disorders) | 2 | 2
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 4
Appendicitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 6
Gangrene (Infections and infestations) | 1 | 2
Diabetic gangrene (Infections and infestations) | 1 | 2
Osteomyelitis (Infections and infestations) | 1 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1
Extradural abscess (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 7
Bronchitis (Infections and infestations) | 1 | 3
Lung infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 3
Urosepsis (Infections and infestations) | 1 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Streptococcal infection (Infections and infestations) | 1 | 0
Streptococcal urinary tract infection (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Gastrointestinal viral infection (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Electrocardiogram ST segment elevation (Investigations) | 1 | 0
Angiogram (Investigations) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 5
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 7 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 2
Cerebral infarction (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 5 | 3
Encephalopathy (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 1 | 1
Central pain syndrome (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 3
Delusion (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Psychogenic seizure (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 6 | 11
Renal failure (Renal and urinary disorders) | 4 | 6
Renal failure chronic (Renal and urinary disorders) | 2 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal infarct (Renal and urinary disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 3 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 0
Coronary revascularisation (Surgical and medical procedures) | 1 | 0
Foot amputation (Surgical and medical procedures) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 3
Accelerated hypertension (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 2 | 0
Circulatory collapse (Vascular disorders) | 1 | 1
Haematoma (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Venous occlusion (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 1
Peripheral ischaemia (Vascular disorders) | 3 | 3
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 2
Femoral artery occlusion (Vascular disorders) | 0 | 2
Intermittent claudication (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 5
Hypotension (Vascular disorders) | 2 | 0
Arteriovenous fistula (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1603) | Fasiglifam 50 mg (N=1601)
Upper respiratory tract infection (Infections and infestations) | 87 | 75
Bronchitis (Infections and infestations) | 45 | 49
Diarrhoea (Gastrointestinal disorders) | 48 | 44
Urinary tract infection (Infections and infestations) | 43 | 35
Nasopharyngitis (Infections and infestations) | 55 | 61
Hypertension (Vascular disorders) | 40 | 42
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 41
Influenza (Infections and infestations) | 37 | 34
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 40
Dizziness (Nervous system disorders) | 30 | 39
Nausea (Gastrointestinal disorders) | 35 | 33
Anaemia (Blood and lymphatic system disorders) | 26 | 33
Headache (Nervous system disorders) | 32 | 41
Sinusitis (Infections and infestations) | 36 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.